CLINICAL TRIAL: NCT05274230
Title: Sustaining Remission From Posttraumatic Stress Disorder (PTSD) Using Tuned Vibroacoustic Stimulation (TVS) Following MDMA-Assisted Psychotherapy
Brief Title: Sustaining Remission From PTSD Using Tuned Vibroacoustic Stimulation (TVS) Following MDMA-Assisted Psychotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Apollo Neuroscience, Inc. (Industry)
Collaborators: The Board of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AN006; 20214600 (Other: WCG IRB)
Record Dates: First submitted 2022-02-18; First posted 2022-03-10 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: remission; PTSD; psychotherapy; MDMA
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a single group study. All participants will receive identical instructions regarding the device and will complete the same survey measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MDMA-Assisted Psychotherapy Participants (Experimental): Participants who have completed the MDMA-Assisted Psychotherapy and consented to be part of this study will use an Apollo Device TVS (10-200 Hz) attached to the subject's wrist or ankle via a commercially available wearable vibration technology can deliver TVS (Transcutaneous Vibratory Stimulation). The intensity will be targeted for the sensory threshold (the level at which the vibration is just noticeable) as this is where the TVS seems to be most effective from prior studies. Similar vibratory stimuli have been demonstrated to be safe in the literature.10-14 The intensity of the vibration will be adjusted to the subjects' comfort and can be controlled by the subject at any time.
  Interventions: Device: Apollo Wearable

INTERVENTIONS:
Device: Apollo Wearable — Participants will be provided with the Apollo wearable device and asked to install the study mobile application on their mobile phone. Participants will use the Apollo for at least 30 minutes after waking up in the morning and at least 30 minutes before bed on the corresponding settings for those times of day. They will be given the Apollo Device TVS (10-200 Hz) to borrow which they will be instructed to wear everyday. They will be asked to continue to wear the device until all study data is collected.
  Other Names: Apollo Neuro

SUMMARY:
The purpose of this research is to examine a wearable device called Apollo that emits gentle vibrations found to benefit mood, energy, and focus. We want to understand how it affects outcomes related to MDMA-assisted psychotherapy for PTSD including depression, anxiety and emotion regulation.

This study will test whether regular use of the Apollo wearable improves rates of sustained symptom remission in PTSD following MDMA-assisted psychotherapy over the course of two years

DETAILED DESCRIPTION:
The study examines the effect of the Apollo wearable on its users after undergoing MDMA-assisted psychotherapy. There will be no study specific modification to the MDMA-assisted psychotherapy that participants receive. All study participants will have previously consented to MAPS MDMA-assisted psychotherapy for PTSD clinical trial before enrolling in this protocol. Once they have been identified as people who have been consented to the MAPS trial regardless of this research, they will be approached about the study, and screened/consented/enrolled accordingly.

Participants will receive the Apollo wearable device via mail upon consenting to participate in this study. They will be provided an instruction manual with guidelines on how to best use the device and will be asked to continue to use the Apollo device in their everyday life following MDMA-assisted psychotherapy.

Participants in the study will be asked to complete monthly online questionnaires for the duration of the two year study.

Please note: this study is not affiliated with the MAPS organization who is running the MDMA-assisted psychotherapy research study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Completion of the MAPS MDMA-Assisted Psychotherapy for PTSD clinical trial (treatment cohort)
* completion of the MAPS MDMA-Assisted Psychotherapy for PTSD clinical trial (placebo cohort)
* enrolled in the MAPS MDMA-Assisted Psychotherapy for PTSD clinical trial, but dropped out

Exclusion Criteria:

* Unable to give adequate informed consent
* Have any current problem which, in the opinion of the investigator might interfere with participation
* Are unable to complete questionnaires written in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Through study completion, an average of two years
  PTSD Checklist for DSM-5 (PCL-5) will be used to measure symptoms of PTSD.
Beck Depression Inventory II (BDI-II) | Through study completion, an average of two years
  Beck Depression Inventory II (BDI-II) will be used to measure symptoms of depression.

SECONDARY OUTCOMES:
World Health Organization Health and Work Performance Questionnaire (HPQ Short form) | Through study completion, an average of two years
  World Health Organization Health and Work Performance Questionnaire (HPQ Short form) will be used to measure work performance.
Alcohol Use Disorders Identification Test (AUDIT) | Through study completion, an average of two years
  Alcohol Use Disorders Identification Test (AUDIT) will be used to measure alcohol use.
Drug Use Disorders Identification Test (DUDIT) | Through study completion, an average of two years
  Drug Use Disorders Identification Test (DUDIT) will be used to measure drug use
Chronic Pain Grade Scale (CPGS) | Through study completion, an average of two years
  Chronic Pain Grade Scale (CPGS) will be used to provide a measure of symptoms of pain. The CPGS is a multidimensional measure that assesses 2 dimensions of overall chronic pain severity: pain intensity and pain-related disability. The 3 subscale scores (characteristic pain intensity, disability score, and the disability points score) are used to classify subjects into 1 of the 5 pain severity grades: grade 0 for no pain, grade I for low disability-low intensity, grade II for low disability-high intensity, grade III for high disability-moderately limiting, and grade IV for high disability-severely limiting.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Tan, MD PhD, Principal Investigator — The Board of Medicine
Locations (1):
- Apollo Neuroscience, Inc., Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Participants who are interested in the study can use the screener link to verify their eligibility — https://apolloneuro.qualtrics.com/jfe/form/SV_5dKbUYhJWJ0B17U